CLINICAL TRIAL: NCT00002987
Title: Minimal Initial Therapy (MIT) for "Early" Supradiaphragmatic Hodgkin's Disease: A Multicenter Randomized Trial of Short Neoadjuvant Chemotherapy (VAPEC-B) Plus Involved Field Radiotherapy (MIT) Versus Mantle Radiotherapy
Brief Title: Combination Chemotherapy Given With Radiation Therapy or Radiation Therapy Alone in Treating Patients With Early-Stage Hodgkin's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065522; MRC-UKLG-LY07; EU-97004
Record Dates: First submitted 1999-11-01; First posted 2004-04-06 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2005-03

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Cyclophosphamide; Doxorubicin; Etoposide; Prednisolone; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: prednisolone
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy plus radiation therapy with radiation therapy alone in treating patients with early-stage Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the recurrence rate and long term survival of patients with early stage Hodgkin's disease given vincristine/doxorubicin/prednisolone/ etoposide/cyclophosphamide/bleomycin (VAPEC-B) chemotherapy and involved field radiation vs mantle radiotherapy.

OUTLINE: This is a randomized multicenter study. Patients are randomized to receive either vincristine/doxorubicin/prednisolone/etoposide/cyclophosphamide/ bleomycin (VAPEC-B) chemotherapy and involved field radiotherapy or mantle radiotherapy only. Patients receiving VAPEC-B are given prednisolone daily on weeks 1-6, doxorubicin IV along with cyclophosphamide IV on week 1, doxorubicin IV and etoposide orally for 5 days on week 3, and vincristine and bleomycin IV on weeks 2 and 4. Involved field radiotherapy is commenced at week 6, within 14 to 21 days of the last chemotherapy treatment. Patients randomized to receive mantle radiotherapy only are given treatments daily for 4 weeks. Patients are followed every 3 months for the first two years, every 4 months for the third year, every 6 months for the fourth and fifth years and annually thereafter.

PROJECTED ACCRUAL: 400 patients will be accrued over 4-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IA or IIA Hodgkin's disease without mediastinal bulk Patients with Hodgkin's disease existing below diaphragm only are not eligible

PATIENT CHARACTERISTICS: Age: 16 to 75 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not HIV positive No prior malignancy other than basal cell carcinoma or cervical intraepithelial neoplasia

PRIOR CONCURRENT THERAPY: No prior treatment

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 1997-01

CONTACTS AND LOCATIONS:
Overall Officials: Michael Williams, MD, Study Chair — Cambridge University Hospitals NHS Foundation Trust
Locations (18):
- Groote Schuur Hospital, Cape Town, Cape Town, South Africa
- United Kingdom (17):
  - University Birmingham, Birmingham, England
  - Bristol Royal Hospital for Sick Children, Bristol, England
  - Bristol Oncology Centre, Bristol, England
  - Addenbrooke's NHS Trust, Cambridge, England
  - Derbyshire Royal Infirmary, Derby, England
  - Cookridge Hospital, Leeds, England
  - University Hospitals of Leicester, Leicester, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Hospital, Northwood, England
  - Norfolk & Norwich Hospital, Norwich, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Royal Marsden Hospital, Sutton, England
  - Southend General Hospital, Westcliff-on-Sea, England
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Preston Hospital, Preston

REFERENCES:
- [Result] Radford JA, Williams MV, Hancock BW, et al.: Minimal initial chemotherapy plus involved field radiotherapy (RT) vs. mantle field RT for clinical stage IA/IIA supra-diaphragmatic Hodgkin's disease (HD). Results of the UK Lymphoma Group LY07 trial. [Abstract] Eur J Haematol 73 (Suppl 65): A-E08, 39, 2004.